CLINICAL TRIAL: NCT00728364
Title: A Case Finding Study for Anderson-Fabry Disease Among Patients With Chronic Kidney Disease Not on Renal Replacement Therapy
Brief Title: Anderson-Fabry Disease in Chronic Kidney Disease Patients Not on Renal Replacement Therapy
Status: Completed | Type: Observational
Sponsor: Klinikum Wels-Grieskirchen (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Manfred Wallner MD, Consultant, Klinikum Wels-Grieskirchen
Other Study IDs: AFD-CKD-Austria-2008
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2012-04

CONDITIONS: Focus of Study: Prevalence of Fabry Disease in CKD Population
Keywords: Anderson Fabry disease; chronic kidney disease; prevalence
MeSH Terms: conditions — Fabry Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Anderson-Fabry disease is a rare X-linked lysosomal storage disorder due to the deficiency of alfa-galactosidase A (AGAL). The subsequent accumulation of glycosphingolipids may lead to to cardiac, renal, and central nervous system impairment as well as premature death. Recently published studies suggest that the true incidence of the disease may be underestimated in certain risk groups, e.g. in patients with chronic kidney disease (CKD).

Therefore, the investigators initiated a multicenter case-finding study in Austria by screening patients with chronic kidney disease not yet on renal replacement therapy. Molecular isoforms of globotriaosylceramide (Gb3), characterized by different chain lengths of their N-acyl residues, will be determined in a urine sample. Characteristic parameters, including the ratio of C24/C18 isoforms will be used for identifying patients liable to have the disease. A positive result will be confirmed by biochemical and genetic testing.

A sample size of 5.000 chronic kidney disease patients is envisaged allowing for detection of 1 to 25 patients with Anderson-Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease KDOQI stage 1-5
* Informed consent

Exclusion Criteria:

* Patients already on renal replacement therapy
* Not willing to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease KDOQI stage 1-5 attending outpatient nephrology clinics in Austria and willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 4353 (Actual)
Dates: Start 2008-10; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Wallner, MD, Principal Investigator — Klinikum Wels-Grieskirchen
Locations (1):
- Klinikum Wels-Grieskirchen, Wels, Upper Austria, Austria

REFERENCES:
- [Result] Kotanko P, Kramar R, Devrnja D, Paschke E, Voigtlander T, Auinger M, Pagliardini S, Spada M, Demmelbauer K, Lorenz M, Hauser AC, Kofler HJ, Lhotta K, Neyer U, Pronai W, Wallner M, Wieser C, Wiesholzer M, Zodl H, Fodinger M, Sunder-Plassmann G. Results of a nationwide screening for Anderson-Fabry disease among dialysis patients. J Am Soc Nephrol. 2004 May;15(5):1323-9. doi: 10.1097/01.asn.0000124671.61963.1e. PMID 15100373